CLINICAL TRIAL: NCT00511030
Title: Assessment of Stability and Ease of Use of a Mail-in Capillary Blood Hemoglobin A!c Sample Kit
Brief Title: Assessment of Stability of Mail-in Capillary Hemoglobin A1c Test Kit
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Uttam Garg, PhD, Children's Mercy Hospital and Clinics
Other Study IDs: 07 06-084E
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Capillary blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the stability of capillary HBA1c blood samples collected by the participant with this kit and mailed to the laboratory at Children's Mercy Hospital.

DETAILED DESCRIPTION:
Participants are given home lab kit for obtaining HbA1c by capillary blood and shipping it to Children's Mercy Hospital and Clinics. They will mail in sample before their next visit and this result will be compared to the HbA1c performed during this visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female diabetic patients ages 1-17 years who have an A1c test drawn within 24 hours
* Participants receiving medical care in the Endocrine Clinic at Children's Mercy Hospital

Exclusion Criteria:

* Not meeting above inclusion criteria

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and females, age 1-17, receiving care in the Endocrine clinic at Children's Mercy Hospital who require HbA1c for standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uttam Garg, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States